CLINICAL TRIAL: NCT01277146
Title: A Phase 1 Dose Escalation Study of OMP-59R5 in Subjects With Solid Tumors
Brief Title: A Dose Escalation Study of OMP-59R5 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59R5-001
Record Dates: First submitted 2011-01-06; First posted 2011-01-14 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors
Keywords: Phase 1; dose escalation; histologically confirmed; malignancy metastatic
MeSH Terms: interventions — tarextumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OMP-59R5 (Experimental)
  Interventions: Drug: OMP-59R5

INTERVENTIONS:
Drug: OMP-59R5 — IV infusion

SUMMARY:
This is an open-label Phase 1 dose escalation study of OMP-59R5 in subjects with previously treated solid tumors for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit. Up to 44 subjects will be enrolled at up to 2 centers. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy. No formal interim analyses will be performed.

Prior to enrollment, subjects will undergo screening to determine study eligibility. Upon enrollment, subjects will receive intravenous (IV) infusions of OMP-59R5 at a assigned dosing schedule for 56 days. After 56 days, subjects will be assessed for disease status. If there is no evidence of disease progression or if the tumor is smaller, then subjects may continue to receive IV infusions of OMP-59R5 every week until disease progression.

Dose escalation will be conducted to determine the maximum tolerated dose (MTD). No dose escalation or reduction will be allowed within a dose cohort. The first 2 subjects enrolled in a cohort will not be treated on the same day. The dose may be administered at any time during the day. Three subjects will be treated at each dose level if no dose-limiting toxicities (DLTs) are observed. The first 2 subjects in each cohort will not be started on OMP-59R5 on the same day. If 1 of 3 subjects experiences a DLT, that dose level will be expanded to 6 subjects. If 2 or more subjects experience a DLT, no further subjects will be dosed at that level and 3 additional subjects will be added to the preceding dose cohort unless 6 subjects have already been treated at that dose level. Subjects will be assessed for DLTs from the time of the first dose through 28 days. Dose escalation for newly enrolled subjects, if appropriate, will occur after all subjects in a cohort have completed their Day 28 DLT assessment. Subjects with stable disease or a response at Day 56 will be allowed to continue to receive weekly doses of OMP-59R5 until disease progression. An additional 14 subjects will be enrolled at the highest dose level that result in <2 of the 6 subjects experiencing a DLT.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed malignancy that is metastatic or unresectable for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit. In addition, subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on CT or MRI.
2. Subjects must have received their last chemotherapy, biologic, or investigational therapy at least 4 weeks prior to enrollment, 6 weeks if the last regimen included BCNU or mitomycin C.
3. Age >18 years
4. ECOG performance status <2 (see Appendix B)
5. Life expectancy of more than 3 months
6. Subjects must have normal organ and marrow function as defined below:

   * Absolute neutrophil count >1000/mL
   * Hemoglobin >9.0 g/dL
   * Platelets >100,000/mL
   * Total bilirubin <1.5 X institutional upper limit of normal (ULN)
   * AST (SGOT) and ALT (SGPT) < 3 X institutional ULN (for subjects with hepatic metastases < 5 X institutional ULN)
   * PT and PTT within 1.5 X institutional ULN
   * Creatinine <1.5 X institutional ULN OR
   * Creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
7. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study, she should inform the Investigator immediately.
8. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Subjects receiving any other investigational agents
2. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants, except for subjects on low molecular weight heparin for DVT/PE prophylaxis. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. New York Heart Association Classification II, III, or IV
10. Subjects with a blood pressure of >140/90 mmHg. The blood pressure must be taken three times 10 minutes apart. Subjects taking antihypertensive medications must be taking ≤ 2 medications to obtain this level of blood pressure control.
11. Subjects with EKG evidence of ischemia or ≥ Grade 2 ventricular arrhythmia, subjects who have a history of acute myocardial infarction within 6 months, or subjects with unstable angina.
12. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease.
13. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease.
14. Subjects with >1 grade 1 diarrhea.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety of OMP-59R5 in subjects with previously treated solid tumors | continuous
  The number of patients experiencing Adverse Events will be reported.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of OMP-59R5 in subjects with previously treated solid tumors | First 8 doses and following treatment termination
  The half-life, volume of distribution, and clearance will be determined
To determine the immunogenicity of OMP-59R5 in subjects with previously treated solid tumors | continuous
  The rate of neutralizing antibodies will be determined
To assess the preliminary efficacy of OMP-59R5 in subjects with previously treated solid tumors | continuous
  The response outcome in patient will be determined

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Principal Investigator — University of Michigan; Anthony W. Tolcher, MD, Principal Investigator — South Texas Accelerated Research Therapeutics, LLC
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- [Derived] Smith DC, Chugh R, Patnaik A, Papadopoulos KP, Wang M, Kapoun AM, Xu L, Dupont J, Stagg RJ, Tolcher A. A phase 1 dose escalation and expansion study of Tarextumab (OMP-59R5) in patients with solid tumors. Invest New Drugs. 2019 Aug;37(4):722-730. doi: 10.1007/s10637-018-0714-6. Epub 2018 Dec 28. PMID 30591982